CLINICAL TRIAL: NCT06242652
Title: A Multicenter, Randomized, Double-blind, Double Dummy，placebo and Positive Controlled，phase II Clinical Study to Evaluate the Efficacy and Safety of 608 in Patients with Ankylosing Spondylitis (AS)
Brief Title: A Study to Evaluate 608 in Patients with Ankylosing Spondylitis (AS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-608-AS-II-01
Record Dates: First submitted 2024-01-22; First posted 2024-02-05 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-02

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 608 Dose A (Experimental): 608 Dose A subcutaneous (SC) injection.
  Interventions: Drug: 608 Dose A
- 608 Dose B (Experimental): 608 Dose B subcutaneous (SC) injection.
  Interventions: Drug: 608 Dose B
- 608 Dose C (Experimental): 608 Dose C subcutaneous (SC) injection.
  Interventions: Drug: 608 Dose C
- Positive control group (Active Comparator): Adalimumab subcutaneous (SC) injection.
  Interventions: Drug: Adalimumab
- Placebo (Placebo Comparator): Placebo subcutaneous (SC) injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 608 Dose A — 608 subcutaneous (SC) injection.
  Other Names: SSGJ-608 Dose A
  Arms: 608 Dose A
Drug: 608 Dose B — 608 subcutaneous (SC) injection.
  Other Names: SSGJ-608 Dose B
  Arms: 608 Dose B
Drug: 608 Dose C — 608 subcutaneous (SC) injection.
  Other Names: SSGJ-608 Dose C
  Arms: 608 Dose C
Drug: Adalimumab — Adalimumab subcutaneous (SC) injection.
  Other Names: Humira
  Arms: Positive control group
Drug: Placebo — Placebo subcutaneous (SC) injection.
  Arms: Placebo

SUMMARY:
This study will evaluate the effect and safety of 608 in patients with AS.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the clinical efficacy, safety and tolerability of 608 compared to placebo and positive drug in patients with AS.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients at least 18 years of age at the time of screening.
2. Participant with a clinical diagnosis of ankylosing spondylitis (AS) and meeting the modified New York criteria for AS.
3. Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score >= 4 and a Patient's Assessment of Total Back Pain score >= 4 based on a 0 - 10 numeric rating scale (NRS) at the Screening and Baseline visits.
4. If entering the study on concomitant NSAIDs for AS, participant must be on stable dose(s) for at least 2 weeks prior to the Baseline visit.

Exclusion Criteria:

1. Patients with other uncontrolled active inflammatory diseases.
2. Clinical laboratory tests and other tests that reveal abnormalities with clinical significance
3. Patients who have active Hepatitis B, Hepatitis C or HIV infections as determined by positive results at Screening.
4. History of cancer.
5. Known or suspected history of immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-02-27 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
The Percentage of Participants Who Achieved an Assessment of Spondylo Arthritis International Society (ASAS) 20 Response. | Week 16.
  Assessment of Spondylo Arthritis International Society criteria (ASAS) consist of 6 domains (4 main and 2 additional assessment domains): 1. Patient's global assessment measured on a NRS; 2. Patient's assessment of back pain, measured on a NRS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions as measured by NRS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) as measured by NRS; 5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
  ASAS 20 response is defined as an improvement of ≥20% and ≥1 unit on a scale of 10 in at least three of the four main domains and no worsening of ≥20% and ≥1 unit on a scale of 10 in the remaining domain. A higher score on the NRS signifies higher severity.

SECONDARY OUTCOMES:
The Percentage of Participants Who Achieved an Assessment of Spondylo Arthritis International Society (ASAS) 40 Response. | Week 16.
  Assessment of Spondylo Arthritis International Society criteria (ASAS) consist of 6 domains (4 main and 2 additional assessment domains): 1. Patient's global assessment measured on a NRS; 2. Patient's assessment of back pain, measured on a NRS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions as measured by NRS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) as measured by NRS; 5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
  ASAS40 response is defined as an improvement of ≥40% and ≥2 units on a scale of 10 in at least three of the four ASAS main domains and no worsening at all in the remaining domain. A higher score on the NRS signifies higher severity.

OTHER OUTCOMES:
608 Concentration in Serum. | Up to 24 Weeks.
  The concentration of 608 in Serum.

CONTACTS AND LOCATIONS:
Locations (1):
- Site 01, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No